CLINICAL TRIAL: NCT01934179
Title: Pilot Study Assessing the Correlation Between Telomere Length and Chemotherapy- Related Toxicity Among Early Stage and Metastatic Colorectal Patients Over the Age of 70
Brief Title: Telomere Length in Predicting Toxicity in Older Patients With Stage III-IV Colorectal Cancer Undergoing Chemotherapy
Status: Terminated | Type: Observational
Why Stopped: Low Accrual Rate
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ERP-GI-049; NCI-2013-01415 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-020 (Other: Fox Chase Cancer Cener); GI-049 (Other: Fox Chase Cancer Center); P30CA006927 (NIH)
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Mucinous Adenocarcinoma of the Colon; Mucinous Adenocarcinoma of the Rectum; Signet Ring Adenocarcinoma of the Colon; Signet Ring Adenocarcinoma of the Rectum; Stage IIIA Colon Cancer; Stage IIIA Rectal Cancer; Stage IIIB Colon Cancer; Stage IIIB Rectal Cancer; Stage IIIC Colon Cancer; Stage IIIC Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-correlative (real-time PCR): Patients undergo blood collection for analysis via real-time PCR at baseline, 3 months, and 6 months.
  Interventions: Other: cytology specimen collection procedure; Other: laboratory biomarker analysis; Other: questionnaire administration

INTERVENTIONS:
Other: cytology specimen collection procedure — Undergo blood sample collection
  Other Names: cytologic sampling
Other: laboratory biomarker analysis — Correlative studies
Other: questionnaire administration — Ancillary studies

SUMMARY:
This pilot research trial studies telomere length in predicting toxicity in older patients with stage III-IV colorectal cancer undergoing chemotherapy. Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in deoxyribonucleic acid (DNA) and predict how well patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the relationship between pre-treatment telomere length (TL) and rate of grade 3 or higher adverse events occurring on front line leucovorin calcium, fluorouracil, and oxaliplatin (FOLFOX)-based chemotherapy among patients over the age of 70 with early stage or metastatic colorectal cancer (CRC).

SECONDARY OBJECTIVES:

I. To evaluate the impact of the FOLFOX-based chemotherapy treatment on peripheral blood lymphocyte telomere length.

II. To evaluate the association between pre-treatment geriatric assessment tools scores, telomere length, and the incidence of chemotherapy related adverse events among older early stage or metastatic CRC patients.

TERTIARY OBJECTIVES:

I. To evaluate the association between pre-treatment levels of serum interleukin-6 (IL-6), C-reactive protein (CRP) and D-dimer and incidence of chemotherapy related adverse events.

II. To evaluate the correlation between pre-treatment telomere length, levels of other biomarkers of aging (IL6, CRP, D-dimer), and rates of adverse events with FOLFOX-based chemotherapy.

OUTLINE:

Patients undergo blood sample collection for analysis via real-time polymerase chain reaction (PCR) at baseline, 3 months, and 6 months.

After completion of study, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Both men and women of all races and ethnic groups are eligible for this trial
* Patients must have histologically or cytologically confirmed adenocarcinoma of the colon or rectum that is stage III or IV and has not been treated with systemic chemotherapy (biopsy of metastatic site not required if primary tumor biopsied and clinical scenario is consistent with metastatic disease)
* Patients must be deemed eligible for systemic chemotherapy with FOLFOX6 +/- bevacizumab at full standard doses
* For patient with metastatic disease, previous adjuvant chemotherapy is allowed as long it was completed at least 12 months prior to study enrollment and did not include oxaliplatin
* Prior radiation therapy is allowed but must have been completed >= 4 weeks prior to study entry
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits, or creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must demonstrate ability to understand and the willingness to sign a written informed consent document
* Patients must demonstrate ability to complete study questionnaires
* Patients must provide written informed consent and Health Insurance Portability and Accountability Act (HIPAA) consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow up
* Male participants with female partners who are of childbearing potential must agree to use an acceptable and effective method of contraception

Exclusion Criteria:

* Patients with metastatic disease who have had adjuvant chemotherapy with oxaliplatin within 12 months of enrollment (single agent fluorouracil [5FU] or capecitabine is allowed) or radiotherapy within 4 weeks prior to entering the study
* Patients with known brain metastases should be excluded from this clinical trial
* Patients with a known history of allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection-requiring intravenous (IV) antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known human immunodeficiency virus (HIV)-positive patients and those with known hepatitis B or C are excluded from the study
* Patients with evidence of other cancer within 5 years, excluding adequately treated basal cell carcinoma of the skin

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09-11 (Actual); Study Completion 2015-09-11 (Actual)

PRIMARY OUTCOMES:
TL | Up to 6 months
  TL will be compared between participants experiencing at least 1 adverse event and those who experience none using the Mann-Whitney test. A type I error of 5% will be used to determine statistical significance.
Incidence of chemotherapy related grade 3 or higher adverse events, graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 6 months
  Variance stabilizing and normalizing transformations will be applied to the data when appropriate. Descriptive statistics for participant characteristics, disease presentation, treatment related toxicity, treatment, duration of chemotherapy use, management of adverse events, and frequency of treatment discontinuation will be tabulated. TL will be compared between participants experiencing at least one adverse event and those who do not experience any adverse event using the Mann-Whitney test. A type I error of 5% will be used to determine statistical significance.

SECONDARY OUTCOMES:
Change in TL after chemotherapy | Baseline to 6 months
  Variance stabilizing and normalizing transformations will be applied to the data as and when appropriate. TL measured at 3 months and at 6 months after chemotherapy treatment will be compared to baseline (pre-treatment) using the Wilcoxon test or the paired t-test as appropriate. A type I error of 5% will be utilized to determine statistical significance. Pre- and post-treatment TL will be summarized using descriptive statistics.

OTHER OUTCOMES:
Association of each geriatric scale, and pro-inflammatory markers to the incidence of chemotherapy related adverse events and TL | Up to 6 months
  Continuous variables will be assessed using the Kruskal-Wallis test or analysis of variance as appropriate and categorical variables will be assessed using Fisher's exact test. Wherever appropriate, Pearson correlation or Spearman's rank correlation will be used to quantify the degree of association between the scales/biomarkers and TL.

CONTACTS AND LOCATIONS:
Overall Officials: Efrat Dotan, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States